CLINICAL TRIAL: NCT01964391
Title: An Open-Label, Multinational, Multicenter, Phase IIIb Study With Subcutaneous Administration of Trastuzumab in Patients With HER2-Positive Early Breast Cancer to Evaluate Patient Satisfaction
Brief Title: A Study of Participant Satisfaction and Safety With Subcutaneously Administered Trastuzumab (Herceptin) in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28851
Record Dates: First submitted 2013-10-08; First posted 2013-10-17 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Doxorubicin; Cyclophosphamide; Paclitaxel; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab (Experimental): In adjuvant setting trastuzumab will be administered in the following treatment regimens: (a) trastuzumab following surgery, chemotherapy (neo-adjuvant or adjuvant) and radiotherapy (if applicable); (b) trastuzumab following adjuvant chemotherapy with doxorubicin and cyclophosphamide, in combination with paclitaxel or docetaxel; (c) trastuzumab in combination with adjuvant chemotherapy consisting of docetaxel and carboplatin. In neo-adjuvant setting, trastuzumab will be administered in combination with neo-adjuvant chemotherapy followed by adjuvant trastuzumab, for locally advanced (including inflammatory) breast cancer or tumors greater than (>) 2 centimeters (cm) in diameter.
  Interventions: Drug: Trastuzumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Docetaxel; Drug: Carboplatin; Drug: Neo-adjuvant chemotherapy

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered subcutaneously at a fixed dose of 600 mg (irrespective of body weight) every 3 weeks for 1 year (adjuvant or neo-adjuvant plus adjuvant therapy).
  Other Names: Herceptin
Drug: Doxorubicin — Doxorubicin will be administered in combination with trastuzumab and cyclophosphamide in the adjuvant setting as per local Product Information and the investigator's discretion.
Drug: Cyclophosphamide — Cyclophosphamide will be administered in combination with trastuzumab and doxorubicin in the adjuvant setting as per local Product Information and the investigator's discretion.
Drug: Paclitaxel — Paclitaxel will be administered in combination with trastuzumab in the adjuvant setting as per local Product Information and the investigator's discretion.
Drug: Docetaxel — Docetaxel will be administered in combination with trastuzumab in the adjuvant setting as per local Product Information and the investigator's discretion.
Drug: Carboplatin — Carboplatin will be administered in combination with trastuzumab and docetaxel in the adjuvant setting as per local Product Information and the investigator's discretion.
Drug: Neo-adjuvant chemotherapy — Neo-adjuvant chemotherapy will be administered according to local guidelines in combination with trastuzumab in the neo-adjuvant setting. The study protocol does not mention any specific neo-adjuvant chemotherapy drug names.

SUMMARY:
This Phase IIIb, open-label, multinational, multicenter study will evaluate the participant's satisfaction and safety with subcutaneously administered trastuzumab in participants with HER2-positive early breast cancer. Participants will receive trastuzumab 600 milligrams (mg) administered subcutaneously every 3 weeks in the adjuvant or neo-adjuvant plus adjuvant setting for 18 cycles (1 year), unless disease progression or unacceptable toxicity occurs. The trastuzumab regimen could include mono- and/or combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hormonal therapy will be allowed as per institutional guidelines
* Prior use of anti-HER2 therapy will be allowed, except for early breast cancer participants in the neo-adjuvant setting
* Left ventricular ejection fraction (LVEF) of greater than or equal to (>=) 55 percent (%) measured by echocardiography (ECHO) or multiple gated acquisition (MUGA) scan prior to first dose of trastuzumab, or, for those who were receiving trastuzumab when beginning the study, documented results within an acceptable limit from a cardiac assessment within 3 months prior to enrollment
* HER2-positive disease immunohistochemistry 3 plus (IHC3+) or in situ hybridization (ISH) positive as determined in a local laboratory that is experienced/certified in HER2-expression testing using an accurate and validated assay
* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast
* No evidence of residual, locally recurrent or metastatic disease after completion of surgery and chemotherapy, or during concurrent chemotherapy (neo-adjuvant or adjuvant)
* Use of concurrent curative radiotherapy will be permitted

Exclusion Criteria:

* History of other malignancy which could affect compliance with the protocol or interpretation of results. Participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma, and participants with other curatively treated malignancies who have been disease-free for at least 5 years, are eligible
* Severe dyspnea at rest or requirement for supplementary oxygen therapy
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab, specifically: history of documented congestive heart failure (CHF), high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), diagnosed poorly controlled hypertension
* Known infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Pregnant or lactating women
* Concurrent enrollment in another clinical trial using an investigational anti-cancer treatment, including hormonal therapy, bisphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin, or a history of severe allergic or immunological reactions, e.g. difficult to control asthma
* Inadequate bone marrow, hepatic or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Participant Satisfaction Questionnaire Score | Week 52
Percentage of Participants with Adverse Events (AEs) | Baseline up to 4.5 years

SECONDARY OUTCOMES:
Healthcare Professional Experience and Satisfaction Questionnaire Score | Week 52
Overall Survival (OS) | Baseline until death from any cause (up to 4.5 years)
Disease-Free Survival (DFS) | Baseline until first documented disease or death, whichever comes first (up to 4.5 years)
  Diagnosis of breast cancer relapse will be made based on routine clinical, radiological and laboratory criteria. Acceptable methods of confirmation of recurrence include radiology, computed tomography (CT) scan, brain scan, ultrasound, or cytology, as per local practice. In case of uncertainty, disease relapse should be confirmed by histological or cytological examination of a suspicious lesion, if possible.
Number of Days on Trastuzumab Treatment | Baseline up to 1 year
Total Daily Dose of Trastuzumab | Baseline up to 1 year
Cumulative Dose of Trastuzumab | Baseline up to 1 year
Duration of Treatment, Follow-up, and Safety Observation | Baseline up to 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Algeria (4):
  - Centre hospitalo-univerisitaire de Rouiba;Service d'oncologie médicale, Algiers
  - Centre Anti Cancer Beau-fraisier;Service d'oncologie médicale, Algiers
  - CHU Annaba; Service d'Oncologie Médicale, Annaba
  - EHS Oncologie Emir Abdelkader Oran; Service d'Oncologie Médicale, Oran
- Morocco (3):
  - Clinique Littoral, Casablanca
  - Centre Hospitalier Universitaire Mohamed VI; Oncologie-Hématologie, Marrakesh
  - Institut National D'oncologie Sidi Med Benabdellah, Rabat
- Saudi Arabia (2):
  - International Medical Center (IMC), Jeddah
  - King Khaled Uni Hospital; Oncology, Riyadh
- Tunisia (4):
  - Abderrahmen Mami Hospital; Medical Oncology department, Aryanah
  - Habib Bourguiba Hospital; Oncology department, Sfax
  - Farhat Hached Hospital; Oncology department, Sousse
  - Institut Salah Azaïz; Service de Médecine Carcinologique, Tunis
- Turkey (Türkiye) (10):
  - Gazi University Medical Faculty; Department of İnternal Medicine, Ankara
  - Akdeniz Univesity Medical Faculty, Antalya
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya University Medical Faculty, Edirne
  - Gaziantep Univ. Med. Fac., Gaziantep
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi, Istanbul
  - Bezmialem Vakif Univ Medical, Istanbul
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Ege University Medical Faculty, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara